CLINICAL TRIAL: NCT07385157
Title: Acceptability and Impact of Ultra-long-term Subcutaneous EEG Monitoring in People With Epilepsy and Intellectual Disability
Brief Title: Ultra-long-term EEG Monitoring in PwID
Status: Active, not recruiting | Type: Observational
Sponsor: University of Plymouth (Other)
Collaborators: Newcastle University (Other); UNEEG Medical A/S (Industry)
Responsible Party: Principal Investigator, Edward Meinert, PhD, Professor of Digital Health and Clinical Artificial Intelligence, University of Plymouth
Other Study IDs: 24NEU030
Record Dates: First submitted 2026-01-05; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Epilepsy; Intellectual Disability, Mild to Moderate
Keywords: Epilepsy; Intellectual Disability; Persons with Mental Disabilities; Electroencephalography; Seizures; Monitoring, Ambulatory
MeSH Terms: conditions — Epilepsy; Intellectual Disability; Seizures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort in people with intellectual disability and epilepsy: The target population of the study will include adult patients who are clinically diagnosed with mild to moderate intellectual disability and epilepsy who are recommended for EEG monitoring by their healthcare professional, their family members or carers, and the clinician responsible for their care.
  Interventions: Device: A minimally-invasive EEG monitoring device

INTERVENTIONS:
Device: A minimally-invasive EEG monitoring device — The minimally-invasive EEG monitoring device (UNEEG Medical's 24/7 EEG SubQ solution) has been CE marked and will be used only in line with its intended use, which includes the population to be investigated in this study. The 2-channel 24/7 EEG SubQ solution is intended for measuring and recording electrical activity of the brain (EEG) through electrodes implanted subcutaneously in the tissue between the skull and the skin. Intended for participants where single location, continuous, ultra-long-term (more than two weeks) EEG recordings are indicated to aid in monitoring and diagnosis of diseases or conditions that alter the EEG. The intended users of the product are males and females, age 18 and above.

SUMMARY:
Many people with intellectual disabilities (PwID) have seizures. Electroencephalography (EEG), which measures the brain's electrical activity, is a key method of diagnosing and assessing seizures but can be difficult and uncomfortable for PwID. UNEEG medical has developed a very small device ('SubQ') that can be put under the skin on a person's head to track their brain activity without staying in the hospital. It has been implanted for 15 months successfully in people with seizures but not in PwID.

The aim of this project is to use learnings from previous co-production work to test how well the device can detect seizures in people with mild to moderate ID and to assess its safety and impact on quality of life and behaviour. The project will also look into carer and clinican experiences using the system and its potential usefulness and cost impact.

Having an accurate means of identifying seizures is particularly important for people with mild to moderate ID because they cannot always tell us about their experiences in a meaningful manner. This means that seizures are more likely to be missed or attributed to behavioural issues.

Healthcare professionals will identify eligible patients to be invited to participate in the study. These patients will be diagnosed with mild to moderate ID, but will have the capacity to consent to take part in the study. The patients who participate in the study will have the UNEEG SubQ device implanted under the skin on their scalp. Ongoing EEG data from the device will be collected and be compared with seizure diaries. The project will also examine any behaviour issues and quality of life using surveys before implantation as well as immediately, 3-months, and 6-months after. The patients, their carers and healthcare professionals will be invited to focus groups to share their experiences with the technology.

ELIGIBILITY:
Patients:

* Adults over 18 years old
* Clinical diagnosis of epilepsy, considered pharmacoresistant
* Clinical diagnosis of mild to moderate ID based on the Diagnostic and Statistical Manual of Mental Disorders (5th ed.; DSM-5; American Psychiatric Association, 2013) and the International Statistical Classfication of Diseases and Related Health Problems (11th ed; ICD-11; World Health Organisation, 2022).Patient has the capacity to consent to take part in the study, and does so
* Able to tolerate the dummy device (device worn for at least 40% of a 1-2 week test period)

Family member / carer:

* Family member/carer is willing to keep a routine seizure diary for the course of the study
* Retrospective seizure diary data available for the proceeding last 6 months
* According to family member, carer, or clinical record, the participant is having at least monthly 'episodes of interest' (it may be unclear whether these are epileptic or behavioural episodes)
* Agree to participate to the study, and support study activities and comply to these

Healthcare professional:

* PwID recommended by their epileptologist for long-term EEG monitoring
* Agree to participate to the study, and support study activities and comply to these

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population of the study will include adult patients who are clinically diagnosed with mild to moderate intellectual disability and epilepsy who are recommended for EEG monitoring by their healthcare professional, their family members or carers, and the clinician responsible for their care.
  Involvement of a participants' family member and/or established carer will be mandatory for the study participation, to safeguard the participants' safety, rights, and well-being throughout the study. A primary carer (family member or professional, depending on the case) for the participant will be involved in the study and answer the questionnaires directed to the carer, participate in feedback consultation with the investigator, handle the device, keep a seizure diary and participate in focus groups to provide research data on behalf of the participant and their own experience.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2024-10-12 (Actual); Primary Completion 2025-11-12 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Device acceptability | At 6 months post-implantation of the device
  The acceptability of the 24/7 SubQ device will be assessed using qualitative data about family members' and carers' perceptions of the patients' experiences with the device. The data will be collected from semi-structured focus groups.
Device adherence | Across 6 months post-implantation of the device
  The adherence to use of UNEEG SubQ device will be assessed using participants' percentage wear time with 24/7 EEG SubQ.
Device usability | At 6 months post-implantation of the device
  The usability of the UNEEG SubQ device will be measured using the average score at 6 months (before explantation) on the System Usability Scale (SUS). The SUS is a 5-point Likert scale 10 items, from strongly disagree (score = 1) to strongly agree (score = 5) [1].

SECONDARY OUTCOMES:
Device safety | From implantation to explantation of the device
  The safety of real-world implementation with 24/7 EEG SubQ Solution in this population will be assessed using the number of adverse events reported during the study period.
Seizure detection accuracy | Across 6 months post-implantation of the device
  The accuracy of seizure detection will be measured by calculating within-participant correlation between seizure counts per month from participant-reported seizure diary and occurrences per month (derived from EEG expert review and annotation of 24/7 EEG SubQ EEG data).
Patients' quality of life | At baseline pre-implantation and post-implantation, and at 3-months and 6 months post-implantation
  The Impact of real-world implementation of the SubQ on quality of life will be measured by the change over time for average Health of the Nation Outcome Scales for people with intellectual disability (HoNOS-ID) scores. The HoNOS-ID includes 18 items, all of which are rated on a 5-point scale from 0 (no problem during the period rated) to 4 (very severe problem) [2].
Patient behaviour | At baseline pre-implantation and post-implantation, and at 3-months and 6 months post-implantation
  The perceived impact of the intervention on patient behaviour will be assessed using the Aberrant Behaviour Checklist (ABC). It includes 58 items, whic are rated on a 4-point scale "from 0 (not at all a problem) to 3 (the problem is severe in degree)" [3].
Satisfaction with the device in daily activities | At 6 months post-implantation of the device
  Patients' satisfaction with the device in daily activities will be assessed using the customised Ease of use scale. This scale consists of 3 items rated on a 1-5 Likert scale, where 1 indicates the most favorable experience (e.g., never limited, very acceptable, never disturbed) and 5 indicates the least favorable experience (e.g., always limited, very unacceptable, always disturbed).
Impact of the device on everyday life | At 6 months post-implantation of the device
  The impact of the device on patients' everyday life will be assessed using a customised questionnaire (named 'Everyday life'). This questionnaire consists of a 5-point rating of overall impact with a free-text explanation of the reasons behind that experience. For the rating, scores range from 1 to 5, where 1 indicates a very positive impact on managing epilepsy in everyday life, and 5 indicates a very negative impact.
Impact of the device on epilepsy management plans | At 3-months and 6 months post-implantation, and every time the clinician initiate a change in the patient's clinical management plan from device implantation untill explantation.
  The impact of the device on epilepsy management plans is measured using a customised questionnaired named 'Epilepsy Management Plan. This questionnaire consists of 5 descriptive items about changes to the epilepsy management plan, reasons for any changes, the role of 24/7 EEG SubQ data in those decisions, the types of adjustments made, and the reasons for not making changes when applicable.
Impact of the device on management of epilepsy | At 3-months and 6 months post-implantation, and every time the clinician initiate a change in the patient's clinical management plan from device implantation untill explantation.
  The impact of the device on management of epilepsy is measured by using a customised questionnaire named 'Management. This questionnaire will be completed by healthcare professionals. It includes three 5-point Likert-scale questions (scored from 1 to 5, where 1 represents a very negative impact or strong disagreement and 5 represents a very positive impact or strong agreement) and two free-text questions about how UNEEG device data influence healthcare professionals' epilepsy management, confidence, and perceptions of patient engagement.
Impact of the device on communication with carers | At 3-months and 6 months post-implantation, and every time the clinician initiate a change in the patient's clinical management plan from device implantation untill explantation.
  The impact of the device on communication with carers about the patient's epilepsy will be assessed using a customised questionnaired named 'Communication'. This questionnaire includes one 5-point Likert-scale question (scored from 1 to 5, where 1 indicates a very negative impact and 5 indicates a very positive impact on the healthcare professional's conversation with the patient's carer) and one free-text question exploring the reasons behind such an impact.
Impact of the device on insights about the patient's epilepsy | At 3-months and 6 months post-implantation, and every time the clinician initiate a change in the patient's clinical management plan from device implantation untill explantation.
  The Impact of the device on insights about the patient's epilepsy is measured using a customised questionnaire named 'Insight'. This questionnaire includes one 5-point Likert-scale question (scored from 1 to 5, where 1 indicates strong disagreement and 5 indicates strong agreement regarding the value of the device data for gaining insight into the patient's epilepsy) and two categorical questions about which epilepsy-related parameters and additional insights beyond standard of care and clinical data were identified or supported by the device data.
Device potential in clinical practice | At 6 months post-implantation of the device
  The potential of the UNEEG device in clinical practice for patients with epilepsy is measured by using a customised questionnaire named 'Potential of 24/7 EEG SubQ'. This questionnaire comprises two 11-point numerical rating questions (scored from 0 to 10, where 0 represents very unsatisfied/very unlikely and 10 represents very satisfied/very likely), five 5-point Likert-scale questions (scored from 1 to 5, where 1 indicates strong disagreement and 5 indicates strong agreement regarding the clinical value and impact of the device), and one free-text question about the perceived potential of the UNEEG device in clinical practice for patients with epilepsy and intellectual disability.
Device deficiency | From device implantation until explantation
  Device deficiencies will be assessed by the number of device deficiencies reported during the study period.

CONTACTS AND LOCATIONS:
Locations (1):
- Cornwall Partnership NHS Foundation Trust, Truro, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Patient identifiable data will not be sold to any other party and will not be shared with any organisation unless they are a partner in the study and have an appropriate information sharing agreement in place.

REFERENCES:
- [Background] [3] Farmer C, Aman MG. Aberrant Behavior Checklist. Encyclopedia of Autism Spectrum Disorders Springer New York; 2020;1-8.
- [Background] [2] Health of Nation Outcome Scales (HoNOS). Royal College of Psychiatrists. 2023. Available from: https://www.rcpsych.ac.uk/improving-care/ccqi/health-ofnation-outcome-scales [accessed May 10, 2024]
- [Background] [1] Brooke J. SUS: a quick and dirty usability scale. ResearchGate. 1995. Nov, [2021-11-21]. https://www.researchgate.net/publication/228593520_SUS_A_quick_and_dirty_usability_scale